CLINICAL TRIAL: NCT00304434
Title: Oseltamivir (Tamiflu) Dosing Strategies for Use During Influenza Prophylaxis (VA01)
Brief Title: Evaluation of Alternative Oseltamivir (Tamiflu) Dosing Strategies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Holodniy, Mark - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: INDA-014-05F
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Influenza
Keywords: Adverse effects; Antiviral; Clinical trial; Oseltamivir; Pharmacokinetics; Probenecid
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Probenecid

ARMS (1):
- 1 (Other)
  Interventions: Drug: Oseltamivir; Drug: Probenecid

INTERVENTIONS:
Drug: Oseltamivir
Drug: Probenecid

SUMMARY:
Objective 1: Determine the safety and toxicity profile of Tamiflu administered in combination with probenecid in healthy adults.Objective 2: Determine the pharmacokinetic profile of Tamiflu and probenecid in healthy adults.

DETAILED DESCRIPTION:
In vitro studies have determined that the 50 % inhibitory concentrations (IC50) of Ro 64-0802 against influenza neuraminidases ranged from 0.3 to 22 nmol/L (0.08 - 0.28 g/L or 0.08 -0.28 ng/mL). IC50 values against influenza strains in cell culture were somewhat higher and more variable ranging from 0.6 to 155 nmol/L (0.17 - 32.8 g/L or 0.17 - 32.8 ng/mL). Tamiflu has also been shown to have in vitro and mouse challenge activity against the H5N1 virus. EC50 values against H5N1 strain replication in Madin Darby canine kidney (MDCK) cells ranged from 7.5-12 M and neuraminidase activity from 7.0-15 nM (IC50 values).

The current U.S. FDA approved recommendations for influenza A and B treatment using oseltamivir suggest a dose of 75mg taken orally twice daily for 5 days at the onset of symptoms or laboratory confirmation of infection. Prophylaxis against influenza A infection for those people exposed to or at high risk for exposure suggests a dose of 75 mg orally taken once daily for up to 6 weeks. No clinical trials in humans infected with or requiring prophylaxis for the H5N1 variant have been performed. Oseltamivir treatment in a human pediatric case of H5N1 influenza pneumonia has been published. Oseltamivir was given late in the course of illness and the child subsequently expired. Several people were given a prophylactic course of oseltamivir after avian influenza (H7N7, H7N3) outbreaks in the Netherlands and in British Columbia, which appeared to be effective in preventing additional human cases.

Clinical trials using oseltamivir for influenza treatment have recently been reviewed. Two phase III placebo controlled, blinded studies were performed in adults, three in geriatric populations, and one in pediatric patients. In general, flu symptoms were decreased by one day or greater in those patients who received Tamiflu compared to placebo. Several prophylaxis studies using oseltamivir have been conducted in healthy unvaccinated adults and have also been recently reviewed. In several trials involving either prophylaxis after household exposure or after exposure in the community have demonstrated that the incidence of influenza was significantly reduced (range 70-90%) in those patients receiving Tamiflu, 75mg orally once daily for 42 days compared to placebo. Side effect profiles in the prophylaxis studies indicate that nausea and vomiting were more commonly found in the Tamiflu arm when compared to placebo. There was no difference in side effect incidence in younger compared to older adult (> 65 years) populations.

ELIGIBILITY:
Inclusion Criteria:

Subjects will include males and non-pregnant females 18 years or older Subjects who can understand the study and potential safety concerns and can sign the informed consent form prior to admission to this study Subjects that are willing to complete all the required assessments, tests and evaluations and able to make all study visits Hemoglobin > 10.0 g/dL for males and > 9.0 g/dL for females; b) Platelet count of > 75,000 / L; c) Absolute neutrophil count > 1000 / L; SGOT and SGPT < than 2.5 times normal upper limit (UL); Serum uric acid WNL; Creatinine < 1.5 times normal upper limit (normal UL 1.5 mg/dL) for the < 65 years of age group and MUST be WNL for the > 65 years of age group; creatinine clearance > 50 mL/min

Exclusion Criteria:

Subjects with a creatinine clearance of < 50 mL/min Subjects who are pregnant or breast feeding females Subjects who are not employing adequate contraception Subjects who are drug or alcohol abusers and in the opinion of the investigator would interfere with subject compliance and safety Subjects who are currently participating in any other clinical research study Any acute serious infection requiring prescription therapy within 14 days prior to Day 1 of the study Subjects who may have or recently been exposed to influenza Subjects with gout, blood dyscrasias, or history of hypersensitivity to sulfonamide drugs Subjects with contraindications to the study medications History of allergic reaction to probenecid Have kidney disease, kidney stones, or poorly functioning kidneys Have active peptic ulcer disease On high dose aspirin or salicylate therapy

Receiving any of the following medications (relative contraindication for probenecid):

Acyclovir, allopurinol, penicillamine, clofibrate, rifampin, methotrexate, zidovudine, theophylline, dapsone, penicillins or cephalosporins, nonsteroidal anti-inflammatory drugs (NSAIDS) such as ibuprofen (Motrin, Advil, Nuprin, others), ketoprofen (Orudis, Oruvail, Orudis KT), diclofenac (Cataflam, Voltaren), etodolac (Lodine), fenoprofen (Nalfon), flurbiprofen (Ansaid), indomethacin (Indocin), ketorolac (Toradol), nabumetone (Relafen), oxaprozin (Daypro), piroxicam (Feldene), sulindac (Clinoril), tolmetin (Tolectin), and naproxen (Aleve, Anaprox, Naprosyn); a sulfa-based medication such as sulfamethoxazole (Bactrim, Septra, Gantanol), sulfasalazine (Azulfidine), sulfinpyrazone (Anturane), sulfisoxazole (Gantrisin), and others; an oral diabetes medicine such as glipizide (Glucotrol), glyburide (Micronase, Diabeta, Glynase), tolbutamide (Orinase), or tolazamide (Tolinase); a barbiturate such as phenobarbital (Luminal, Solfoton), amobarbital (Amytal), secobarbital (Seconal), and others; or a benzodiazepine (used to treat anxiety and panic disorders and to induce sleep) such as alprazolam (Xanax), diazepam (Valium), lorazepam (Ativan), temazepam (Restoril), chlordiazepoxide (Librium), clonazepam (Klonopin), clorazepate (Tranxene), oxazepam (Serax), estazolam (ProSom), flurazepam (Dalmane), quazepam (Doral), or triazolam (Halcion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine whether the combination of oseltamivir and probenecid result in equivalent blood plasma concentrations compared to oseltamivir given alone | 15 days

SECONDARY OUTCOMES:
The safety of combining oseltamivir and probenecid

CONTACTS AND LOCATIONS:
Overall Officials: Mark Holodniy, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Result] He G, Massarella J, Ward P. Clinical pharmacokinetics of the prodrug oseltamivir and its active metabolite Ro 64-0802. Clin Pharmacokinet. 1999 Dec;37(6):471-84. doi: 10.2165/00003088-199937060-00003. PMID 10628898
- [Result] Massarella JW, He GZ, Dorr A, Nieforth K, Ward P, Brown A. The pharmacokinetics and tolerability of the oral neuraminidase inhibitor oseltamivir (Ro 64-0796/GS4104) in healthy adult and elderly volunteers. J Clin Pharmacol. 2000 Aug;40(8):836-43. doi: 10.1177/00912700022009567. PMID 10934667
- [Result] Hill G, Cihlar T, Oo C, Ho ES, Prior K, Wiltshire H, Barrett J, Liu B, Ward P. The anti-influenza drug oseltamivir exhibits low potential to induce pharmacokinetic drug interactions via renal secretion-correlation of in vivo and in vitro studies. Drug Metab Dispos. 2002 Jan;30(1):13-9. doi: 10.1124/dmd.30.1.13. PMID 11744606
- [Result] Holodniy M, Penzak SR, Straight TM, Davey RT, Lee KK, Goetz MB, Raisch DW, Cunningham F, Lin ET, Olivo N, Deyton LR. Pharmacokinetics and tolerability of oseltamivir combined with probenecid. Antimicrob Agents Chemother. 2008 Sep;52(9):3013-21. doi: 10.1128/AAC.00047-08. Epub 2008 Jun 16. PMID 18559644
- [Result] Raisch DW, Straight TM, Holodniy M. Thrombocytopenia from combination treatment with oseltamivir and probenecid: case report, MedWatch data summary, and review of the literature. Pharmacotherapy. 2009 Aug;29(8):988-92. doi: 10.1592/phco.29.8.988. PMID 19637952